CLINICAL TRIAL: NCT04304911
Title: Implementation, Effficacy and Cost-effective Study of the Unified Protocol in Blended Format for Transdiagnostic Treatment of Emotional Disorders in the Spanish National Health System
Brief Title: UP in Blended Format for Transdiagnostic Treatment of Emotional Disorders in the Spanish National Health System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IPES/PI20/00697
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Emotional Disorder; Anxiety Disorders; Depressive Disorder
Keywords: Emotional Disorder; Unified Protocol; Public health; Transdiagnostic approach
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: All consecutive patients with emotional disorders attending any of the collaborating centers will be asked to participate in the present study. Once inclusion criteria are met, each patient will be randomly assigned to one of the two experimental groups: Treatment as Usual (TAU) or UP-APP. Randomization will be performed by a researcher unrelated to the study using a computer-generated sequence (Randomizer). Randomization will be stratified according to the severity of the primary measures of depression and anxiety, using the recommended cutoff in the manuals. Stratification will be made to ensure a comparable proportion of severely depressed and anxious individuals in each group. For each subgroup (i.e., severe or less severe depression and/or anxiety), participants will be randomly assigned to the UP-APP or to TAU.
Who Masked: Participant
Masking Description: Patients (participants) will know the treatment they have been assigned to, but they will not know whether that treatment is considered TAU or experimental (UP-APP). Healthcare professionals and researchers will know the condition each patient has been assigned to (mandatory to provide a given type of intervention).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UP in blended format (Experimental): Clinicians will follow the UP therapist manual, 2nd edition, recently translated by Osma and Crespo (13,14). The same contents through a digital material (video and audio) will be integrated in the UP-APP. The program can be developed in a range of 12 to 16 sessions. The UP includes 8 modules
  Interventions: Behavioral: Blended intervention (UP-APP)
- Treatment as usual (TAU) (Active Comparator): Cognitive Behavioral Therapy in individual format is the treatment of choice (TAU) by psychologists and psychiatrists at the collaborating Public Mental Health Centers and Primary Care Centers, together with pharmacological treatment (i.e., antidepressants and / or anxiolytics).
  Interventions: Behavioral: Cognitive Behavioral Therapy (TAU)

INTERVENTIONS:
Behavioral: Blended intervention (UP-APP) — Unified Protocol (UP) for transdiagnostic treatment of EDs in the blended intervention (UP-APP)
  Arms: UP in blended format
Behavioral: Cognitive Behavioral Therapy (TAU) — TAU group that carries out Cognitive Behavioral Therapy in an individual format
  Arms: Treatment as usual (TAU)

SUMMARY:
The present randomized, controlled trial will compare the efficacy, cost-effectiveness, and implementation characteristics of a blended intervention based on the Unified Protocol (UP) for transdiagnostic treatment of emotional disorders against the treatment as usual in a sample of patients with emotional disorders in the Spanish National Health System.

DETAILED DESCRIPTION:
Emotional disorders (EDs;including anxiety disorders, unipolar mood disorders, and related disorders) are the most prevalent mental disorders in the general population. In Spain, anxiety disorders and mood disorders affect approximately two million (4.1%) and two and half million (5.2%) individuals, respectively. As a result of their prevalence in the society, EDs have become an alarming health problem due to their associate costs. These disorders have a direct cost of 22.000 million euros (500 euros per capita and year). The total expense of these disorders entails 2.2% of the Gross Domestic Product in Spain. Due to the excessive demand for treatment, mental health services of our National Health System (NHS) are collapsed with large waiting lists, which results in a great difficulty to dedicate the recommended time to attend patients who require psychological treatment. Therefore, it is needed to find solutions for the effective and cost-effective treatment of EDs in our NHS. In the last years, several solutions have been proposed to alleviate this important health problem.

The general objective of this project is to contribute to the dissemination of evidence-based psychological treatments in our Public National Health System for the most prevalent mental disorders in our society, emotional disorders (EDs). The investigators will study the efficacy, cost-effectiveness, and implementation characteristics (acceptability, usability, and utility) of a blended intervention which will enhance face-to-face treatment by incorporating an app-based intervention onsite treatment. Based on the most recent clinical advances in the treatment of EDs, the investigators will use the Unified Protocol (UP) for transdiagnostic treatment of EDs in the blended intervention (UP-APP). The investigators hypothesize that the blended intervention will be superior to the treatment as usual (face-to-face, specific-disorder treatment) because patients in the UP-APP condition will continue working with the app at home between sessions. In sum, this project is composed of three connected studies: a validation study in a clinical sample of patients with EDs, two pilot studies to help develop the app based on the UP principles, and a multicenter, randomized and controlled clinical trial that will be conducted by 12 clinical psychologist working in 8 different provinces in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Principal diagnosis of Emotional disorder (Evaluated by MINI interview)
* The patient is over 18 years of age
* The patient is fluent in the language in which the therapy is performed (Spanish in the present study)
* To have a Smartphone
* Patients taking pharmacological treatment for their ED will be asked to maintain the same dosages and medications for at least 3 months prior to enrolling in the study and during the whole treatment
* The patient signs the informed consent form.

Exclusion Criteria:

* The patient presents a severe condition that would require to be prioritized for treatment, these include a severe mental disorder (bipolar disorder, schizophrenia, or an organic mental disorder), suicide risk at the time of assessment, or substance use in the last three months
* The patient has previously received 8 or more sessions of psychological treatment with clear and identifiable Cognitive behavioral therapy (CBT) principles within the past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Overall Depression Severity and Impairment Scale (ODSIS) | Up to 12 months
  Consist of five items that evaluate the frequency and the intensity of depressive symptoms and their interference with the person's work or school life and social life. The total score range from 0 to 20 and responses use a 5-point Likert scale ranging from 0 to 4.
Overall Anxiety Severity and Impairment Scale (OASIS) | Up to 12 months
  The scale presents five items. These items are related with the frequency and intensity of anxiety symptoms and their interference with the person's work or school life and with social life. All items are rated on a 5-point Likert scale ranging from 0 (I didn't feel anxious) to 4 (Constant anxiety).
Anxiety and Related Disorders Interview Schedule for DSM-5 (ADIS-V) | Enrolment and Up to 12 months
  Diagnostic interview

SECONDARY OUTCOMES:
The Multidimensional Emotional Disorder Inventory (MEDI) | Up to 12 months
  A self-report measure that includes only 49 items and enables to quickly assess the main transdiagnostic dimensions of Emotional disorders
Health-related quality of life (EuroQol-5D) | Up to 12 months
  Evaluation through 5 items of quality of life.
Adaptation of Client Satisfaction Questionnaire [CSQ-8] | Up to 12 months
  An adaptation of 13 items that measures quality of the intervention and its components, discomfort experienced during treatment and the experience of participating in a blended format.
Five Facet Mindfulness Questionnaire (FFMQ) | Up to 12 months
  Is a 39-item questionnaire that measures five facets of mindfulness. responses use a 5-point Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true)
Emotion Regulation Questionnaire (ERQ) | Up to 12 months
  Consists of 10 items covering two factors: Cognitive Reappraisal (six items) and Expressive Suppression (four items). Items are rated on a 7-point Likert scale ranging from ''Strongly disagree'' to ''Strongly agree'
Difficulties in Emotion Regulation Scale (DERS) | Up to 12 months
  Consists of 36-item of six facets of emotion regulation. Items are rated on a scale of 1 ("almost never [0-10%]") to 5 ("almost always [91-100%]"). Higher scores indicate more difficulty in emotion regulation
Credibility/Expectancy Questionnaire (CEQ) | Up to 12 months
  The CEQ consists of six items scored on a scale of 1 to 9 and measures treatment expectancy and credibility of justification for use in clinical outcome studies.
System Usability Scale (SUS) | Up to 12 months
  Composed of 10 statements that are scored on a 5-point scale of strength of agreement [0-100]
Client Service Receipt Inventory (CSRI) | Up to 12 months
  Evaluate the emergency service (total visits), general medical inpatient hospital admissions (total days); outpatient health care services (total visits to general practitioner, nurse, social worker, psychologist, and other community health care professionals).
Working Alliance Inventory-Short (WAI-S) | During psychological treatment
  Evaluate the therapeutic or working alliance
Quality-adjusted Life Years (QALYs) | Up to 12 months
  Measure of disease burden, including both the quality and the quantity of life lived. It is used in economic evaluation to assess the value of medical interventions.
UP-APP outcomes | During psychological treatment
  Number and time of use of the UP-APP, videos viewed and exercises completed
Evaluation of the UP-APP | Up to 12 months
  16 items that evaluate the opinion about the app's aesthetics, handling and components
Evaluation questionnaire of the Unified Protocol (UP) modules | Up to 12 months
  Consists of 7 items that evaluate the usefulness of the program to improve emotional regulation and the usefulness of each of the skills that are worked on in the different UP modules

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Osma, Ph.D, Principal Investigator — Instituto de Investigación Sanitaria de Aragón, Universidad de Zaragoza
Locations (1):
- Hospital Comarcal de Vinaròs, Vinaròs, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
Under request

REFERENCES:
- [Derived] Martinez-Garcia L, Schaeuffele C, Peris-Baquero O, Torres Alfosea MA, Osma J. Acceptability and preliminary effectiveness of the Unified Protocol in blended format in the Spanish public mental health system: Results from a Pilot Randomized Controlled Trial. Psychother Res. 2025 Aug 12:1-18. doi: 10.1080/10503307.2025.2541707. Online ahead of print. PMID 40792553
- [Derived] Osma J, Martinez-Garcia L, Peris-Baquero O, Navarro-Haro MV, Gonzalez-Perez A, Suso-Ribera C. Implementation, efficacy and cost effectiveness of the unified protocol in a blended format for the transdiagnostic treatment of emotional disorders: a study protocol for a multicentre, randomised, superiority controlled trial in the Spanish National Health System. BMJ Open. 2021 Dec 31;11(12):e054286. doi: 10.1136/bmjopen-2021-054286. PMID 34972770
- See also: Related Info — https://www.iisaragon.es/grupos-de-investigacion/neurociencia-salud-mental-y-organos-de-los-sentidos/giis082-investigacion-en-personalidad-emocion-y-salud-ipes/
- See also: Related Info — https://www.alianzaeditorial.es/libro/manuales/aplicaciones-del-protocolo-unificado-para-el-tratamiento-transdiagnostico-de-la-disregulacion-emocional-jorge-osma-9788491817260/
- See also: Related Info — https://www.alianzaeditorial.es/libro/manuales/protocolo-unificado-para-el-tratamiento-transdiagnostico-de-los-trastornos-emocionales-manual-del-terapeuta-david-h-barlow-9788491814795/
- See also: Related Info — https://www.alianzaeditorial.es/libro/manuales/protocolo-unificado-para-el-tratamiento-transdiagnostico-de-los-trastornos-emocionales-manual-del-paciente-david-h-barlow-9788491814818/